CLINICAL TRIAL: NCT07360210
Title: Muscle Damage of the TFL (Tensor Fascia Latae) During Total Hip Arthroplasty (THA) Through Direct Anterior Approach (DAA), Evaluation of the Correlation With Short Term Functional Results
Brief Title: Muscle Damage of the TFL (Tensor Fascia Latae) During Total Hip Arthroplasty (THA) Through Direct Anterior Approach (DAA)
Acronym: TFL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2024/83
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Hip Joint; Surgery; Arthroplasty; Replacement; Surgical Wound; Muscle Injury; Fascia Lata
Keywords: TFL damage; Total Hip Arthroplasty through Direct Anterior Approach
MeSH Terms: conditions — Surgical Wound | interventions — Data Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Usual surgical procedure (Other): Patient with usual surgical procedure : Total Hip Arthroplasty through Direct Anterior Approach
  Interventions: Other: Data collection and self-administered questionnaire

INTERVENTIONS:
Other: Data collection and self-administered questionnaire — Data collection and self-administered questionnaire (HHS and SF-36)

SUMMARY:
Direct Anterior Approach (DAA) is known to cause damage to the TFL during the surgical approach, the point of this study is to evaluate the impact between the severity of the per operative TFL damage and the functional short term results.

DETAILED DESCRIPTION:
Total hip arthroplasty is one of the most frequent surgical procedure and it has changed the approach of hip arthrosis. There are a few surgical approaches frequently used : posterolateral approach, anterolateral approach and the direct anterior approach. It has been previously shown that the DAA is causing less muscle damage than the other surgical approaches, the anterior interval is considered as internervous and intermuscular muscle-sparing technique. However, several reports have proved that the DAA was also associated with muscle damage, particularly to the tensor fascia lata during the exposition with the instruments.

The purpose of this study is to determinate the correlation between the severity of muscle damage during surgery and the functional post operative short and medium term results. We underwent grading visible muscle damage during surgery after implant positioning by a grading system in 5 stages from 0 (intact or a few fibers) to 4 (more than 75% of muscle damage). Functional results were established by Harris Hip Score at 6 weeks and 6 months follow up.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 years old),
* patient undergoing primary Total Hip Arthroplasty through Direct Anterior Approach for osteoarthritis

Exclusion Criteria:

* hip dysplasia
* leg length discrepancy greater than 2cm
* history of homolateral hip surgery
* neuromuscular pathology
* patients declining the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between post operative functional results and TFL muscle damage | week 6
  Correlation between :
  * short term post operative functional results, evaluated by Harris Hip score at 6 weeks. Harris Hip score has 10 items with several propositions per each item and total score from 2 to 100 , and
  * TFL muscle damage grade during surgery evaluated with ATHLAS classification : score 0 (intact or few fibres), 1 (0-25% of fibres), 2 (25-50%), 3 (50-75%) et 4 (>75%)

SECONDARY OUTCOMES:
Harris Hip score 6 months | 6 months
  Result of Harris Hip score at 6 months Harris Hip score has 10 items with several propositions per each item and total score from 2 to 100 ,
Quality of life scale | 6 weeks, 6 months
  Evolution of SF-36 questionnaire score between 6 weeks and 6 months after total hip arthroplasty

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Bordeaux, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux